CLINICAL TRIAL: NCT00608101
Title: Hypoglycemia Associated Autonomic Failure in Type 1 DM, Question 1
Brief Title: Hypoglycemia Associated Autonomic Failure in Type 1 Diabetes Mellitus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Steve Davis, Department Chair, Vanderbilt University
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: IRB #040907-HAAF in T1DM, Q1; R01DK069803-03 (NIH)
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes
Keywords: hypoglycemia; exercise; corticosteroids
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Motor Activity | interventions — Fludrocortisone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Day 1 hyperinsulinemic euglycemic clamps with either 0.2 mg fludrocortisone, 0.75 mg Dexamethasone, or both given orally before each morning and afternoon clamp. Day 2 hyperinsulinemic hypoglycemic glucose clamp.
  Interventions: Drug: Fludrocortisone
- 2 (Experimental): Fludrocortisone will be administered in doses of 0.05mg, 0.1mg and 0.2 mg form at the start of each clamp period on day 1. Dexamethasone will be administered orally in the doses of 0.18 mg, 0.375mg and 0.75mg doses. The combination of the 0.05mg fludrocortisone and 0.18mg dexamethasone and 0.1mg of fludrocortisone and 0.375 mg doses will be administered at the start of each day 1 clamp period. Day 2 90 minutes of moderate exercise.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Fludrocortisone — Oral Fludrocortisone 0.2 mg x 2 prior to each experimental period on Day 1
  Arms: 1
Drug: Dexamethasone — Oral Dexamethasone 0.75 mg x 2 administered prior to each experimental period on Day 1
  Arms: 2

SUMMARY:
The purpose of this study is to determine what corticosteroid receptor (and the dose of) is responsible for cortisol inducing hypoglycemia associated autonomic dysfunction in Type 1 DM. Specifically, we aim to determine whether stimulating the type 1 corticosteroid receptor (via fludrocortisone), the type 2 corticosteroid receptor (via dexamethasone), or both causes hypoglycemia associated autonomic dysfunction in Type 1 DM.

ELIGIBILITY:
Inclusion Criteria:

* 16 (8 males, 8 females) Type 1 diabetic patients aged 18-45 yr.
* HbA1c > 7.0%
* Had diabetes for 2-15 years
* No clinical evidence of diabetic tissue complications
* 16 (8 males, 8 females) Healthy volunteers aged 18-45 yrs.
* Body mass index < 27kg · m-2

Exclusion Criteria:

* Prior or current history of poor health
* Abnormal results following blood and physical examination
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
catecholamines | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — Vanderbilt University